CLINICAL TRIAL: NCT01639508
Title: A Phase II Study of Cabozantinib in Patients With RET Fusion-Positive Advanced Non-Small Cell Lung Cancer and Those With Other Genotypes: ROS1 or NTRK Fusions or Increased MET or AXL Activity
Brief Title: Cabozantinib in Patients With RET Fusion-Positive Advanced Non-Small Cell Lung Cancer and Those With Other Genotypes: ROS1 or NTRK Fusions or Increased MET or AXL Activity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-097
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung; XL184 (CABOZANTINIB); KIF5B/RET Positive; RET Fusion Positive; 12-097; Genotypes: ROS1 or NTRK Fusions or Increased MET or AXL Activity
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cabozantinib

ARMS (1):
- Cabozantinib (Experimental): This will be a single-institution, open label, two-stage, single agent trial of cabozantinib in patients with advanced NSCLCs.atients in GROUP A will have tumors with a RET fusion. Patients in GROUP B will have tumors with an NTRK fusion, or MET or AXL overexpression, amplication, or mutatation. Patients in GROUP C will have tumors with a ROS1 fusion. Patients in GROUP D will have tumors with a RET fusion and have progressed on a selective RET TKI.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Patients will receive cabozantinib at an initial dose of 60 mg orally daily. The drug is taken continuously over a period of 28 days (4 weeks), which constitutes one treatment cycle. Dose modifications for drug toxicity are permitted as per a prescribed algorithm. During the Treatment Period subjects will receive cabozantinib until either disease progression, the occurrence of unacceptable drug-related toxicity or for other reason(s) for subject withdrawal.

SUMMARY:
The purpose of this phase II study is to find out what effects cabozantinib (XL184) has, good and/or bad, in patients whose tumors one of the following gene changes RET, ROS1, or NTRK fusion, or increased MET or AXL activity.

A phase II study looks at how effective a medication is at treating a specific type of cancer and collects information on the side effects of the study treatment.

RET, ROS1, or NTRK fusion or increased MET or AXL activity gene leads to lung cancer cell growth. Cabozantinib is an oral medicine that inhibits of RET, ROS1, NTRK, MET, and AXL. In addition, this drug interferes with other cell pathways that also cause cancer cells to grow, form new blood vessels, and spread to other organs of the body. The goal of using cabozantinib is to shrink the cancer and to prevent it from growing

Cabozantinib has been studied and shown to cause cancer shrinkage in other cancers such as medullary thyroid cancer and prostate cancer. We thus have a good idea of what side-effects it causes and can anticipate them.

ELIGIBILITY:
Inclusion Criteria:

A subject must fully meet all of the following criteria to be eligible for the study:

1. The subject has a pathologic diagnosis of non-small cell lung carcinoma that is metastatic or unresectable.
2. Documented presence:

   1. Group A: KIF5B/RET or related variant RET fusions.
   2. Group B: any of the following aberrations

      ii. NTRK fusion iii. MET overexpression, amplification, or mutation iv. AXL overexpression, amplification, or mutation
   3. Group C: ROS1 fusion
   4. GROUP D: RET-fusion post-progression on selective RET inhibitor
3. The subject is ≥ 18 years old on the day of consent.
4. Measurable Disease by RECIST1.1
5. The subject has a Karnofsky performance status of > 70%.
6. The subject has organ and marrow function and laboratory values as follows:

   1. Absolute neutrophil count (ANC) ≥ 1500/mm3 without colony stimulating factor support
   2. Platelets ≥ 100,000/mm3 Hemoglobin ≥ 9 g/dL
   3. Bilirubin ≤ 1.5 × the upper limit of normal (ULN). For subjects with known Gilbert's . disease, bilirubin ≤ 3.0 mg/dL
   4. Serum creatinine ≤ 1.5 × ULN or creatinine clearance (CrCl) ≥ 30 mL/min. For creatinine clearance estimation, the Cockcroft and Gault equation should be used:

      Male: CrCl (mL/min) = (140 - age) × wt (kg) / (serum creatinine × 72) Female:

      Multiply above result by 0.85
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)

      ≤ 3.0 × ULN if no liver involvement, or ≤ 5 × ULN with liver involvement
   6. Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (113.2 mg/mmol) creatinine or 24-hr urine protein of < 1 g
   7. Serum phosphorus, magnesium, and potassium ≥ LLN after adequate supplementation if necessary
   8. The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document. Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (eg, male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control. Women of childbearing potential must have a negative pregnancy test at screening.
   9. Women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal.
   10. Postmenopause is defined as amenorrhea ≥ 12 consecutive months. Note:

women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression or any other reversible reason.

Exclusion Criteria:

1. Any type of systemic anticancer agent (including investigational) within 3 weeks of first dose of study treatment, or within 5 half-lives of the agent whichever is shorter. Subjects on LHRH or GnRH agonists may be maintained on these agents.
2. Prior treatment with cabozantinib
3. Radiation therapy for bone or brain metastasis within 2 weeks, any other external radiation therapy within 4 weeks of first dose of study drug. Systemic treatment with radionuclides within 4weeks. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
4. The subject has not recovered to baseline or CTCAE ≤ Grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant AEs.
5. Known uncontrolled symptomatic brain metastases or cranial epidural disease; subjects previously treated and on stable dose of corticosteroids and/or anticonvulsants for >10 days, or not requiring such medications, are eligible. Baseline brain scans are not required to confirm eligibility.

   Radiation therapy for bone or brain metastases within 2 weeks before first dose of study drug; or any other external radiation therapy or systemic treatment with radionuclides within 4 weeks before first dose of study drug. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
6. The subject requires concomitant treatment, in therapeutic doses, unless deemed clinically unsafe to discontinue, with anticoagulants such as warfarin or warfarin-related agents, unfractionated heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (eg, clopidogrel). Low dose aspirin (≤ 100 mg/day), low-dose warfarin (≤ 1 mg/day) are permitted. Both prophylactic and/or treatment dose low molecular weight (fractionated) heparin (LMWH) are permitted and are the preferred agents to administer.
7. The subject has experienced any of the following within 3 months before the first dose of study treatment:

   * clinically-significant hematemesis or gastrointestinal bleeding
   * Clinically-significant hemoptysis of ≥ 0.5 teaspoon (2.5ml) of red blood c. any other signs indicative of pulmonary hemorrhage
8. The subject has radiographic evidence of cavitating pulmonary lesion(s)
9. The subject has tumor in contact with invading major blood vessels
10. The subject has any evidence of an endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib.
11. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    * Cardiovascular disorders including Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening

      * Concurrent uncontrolled hypertension defined as sustained BP ≥ 150 mm Hg systolic, or ≥ 90 mm Hg diastolic despite optimal antihypertensive treatment (Note: If there is any BP measurement that is performed within the screening period that is < 150 mm Hg systolic and <90 mm Hg diastolic, then BP does not meet definition of sustained.)

        ---- Any congenital history of long QT syndrome.
      * Any of the following within 6 months before the first dose of study treatment:

        * unstable angina pectoris
        * clinically-significant cardiac arrhythmias
        * stroke (including TIA, or other ischemic event) myocardial infarction
        * thromboembolic event requiring therapeutic anticoagulation except if anticoagulation is as stipulated in Exclusion Criterium #6. (Note: subjects with a venous filter (e.g. vena cava filter) are not eligible for this study)
    * Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

      * Any of the following within 28 days before the first dose of study treatmentF

        * intra-abdominal tumor/metastases invading GI mucosa (malignant abdominal ascites does not constitute mucosal invasion)
        * active peptic ulcer disease,
        * inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
        * malabsorption syndrome
      * Any of the following within 6 months before the first dose of study treatment:

        * history of abdominal fistula
        * gastrointestinal perforation
        * bowel obstruction or gastric outlet obstruction
        * intra-abdominal abscess. Note: Complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more that 6 months ago. GI surgery (particularly when associated with delayed or incomplete healing) within 28 days. Note: Complete healing following abdominal surgery must be confirmed prior to initiating treatment with cabozantinib even if surgery occurred more that 28 days ago.
    * Other disorders associated with a high risk of fistula formation including PEG tube placement within 3 months before the first dose of study therapy or concurrent evidence of intraluminal tumor involving the trachea and esophagus.
    * Other clinically significant disorders such as:

      * active infection requiring systemic treatment within 28 days before the first dose of study treatment
      * serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
      * history of organ transplant
      * concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment
      * Major surgery (eg, thoracotomy, removal or biopsy of brain metastasis) within 3 months before Week 1 Day 1. Complete wound healing from major surgery must have occurred 1 month before Week 1 Day 1 and from minor surgery (eg, simple excision, tooth extraction) at least 10 days before Week 1 Day 1. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
      * history of major surgery as follows:
12. The subject is unable to swallow tablets
13. The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms 14 days before Week 1 Day 1
14. The subject is pregnant or breastfeeding.
15. The subject has a previously identified allergy or hypersensitivity to components of the study treatment formulation.
16. The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.
17. Uncontrolled concurrent malignancy that would limit assessment of efficacy of cabozantinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2012-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) (Group A) | 12 weeks
  by RECIST v1.1 criteria to cabozantinib in patients with advanced NSCLC who have tested positive for RET Fusion
objective response rate (ORR) (Group B) | 12 weeks
  by RECIST v1.1 criteria to cabozantinib in patients with advanced NSCLC whose tumors test positive for a ROS1 or NTRK fusion or MET or AXL overexpression, amplification, or mutation.

SECONDARY OUTCOMES:
progression-free survival (PFS) (Group A) | 3 years
  Progression-free (PFS) and overall survival (OS) will be calculated using Kaplan-Meyer estimators starting from the time of treatment initiation. For PFS, patients alive without evidence of progression at the end of the study will be censored at the time of the last available follow-up. For OS, patients alive at the end of the study will be censored at the time of the last available follow-up.
overall survival (OS) (Group A) | 3 years
  Progression-free (PFS) and overall survival (OS) will be calculated using Kaplan-Meyer estimators starting from the time of treatment initiation. For PFS, patients alive without evidence of progression at the end of the study will be censored at the time of the last available follow-up. For OS, patients alive at the end of the study will be censored at the time of the last available follow-up.
safety (Group A, B, C & D) | 3 years
  Observed toxicities will be individually tabulated according to CTCAE version 4.0 and summarized using descriptive statistics.
progression-free survival (PFS) (Group B, C & D) | 3 years
  Progression-free (PFS) and overall survival (OS) will be calculated using Kaplan-Meyer estimators starting from the time of treatment initiation. For PFS, patients alive without evidence of progression at the end of the study will be censored at the time of the last available follow-up. For OS, patients alive at the end of the study will be censored at the time of the last available follow-up with advanced NSCLCs whose tumors test positive for a ROS1 or NTRK fusion or MET or AXL overexpression or amplification who were treated with cabozantinib.
overall survival (OS) (Group B, C & D) | 3 years
  Progression-free (PFS) and overall survival (OS) will be calculated using Kaplan-Meyer estimators starting from the time of treatment initiation. For PFS, patients alive without evidence of progression at the end of the study will be censored at the time of the last available follow-up. For OS, patients alive at the end of the study will be censored at the time of the last available follow-up with advanced NSCLCs whose tumors test positive for a ROS1 or NTRK fusion or MET or AXL overexpression or amplification who were treated with cabozantinib.

OTHER OUTCOMES:
objective response rate (ORR) (Group D) | 12 weeks
  by RECIST v1.1 criteria to cabozantinib in patients with advanced NSCLC who have tested positive for RET Fusion

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Drilon, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Drilon A, Rekhtman N, Arcila M, Wang L, Ni A, Albano M, Van Voorthuysen M, Somwar R, Smith RS, Montecalvo J, Plodkowski A, Ginsberg MS, Riely GJ, Rudin CM, Ladanyi M, Kris MG. Cabozantinib in patients with advanced RET-rearranged non-small-cell lung cancer: an open-label, single-centre, phase 2, single-arm trial. Lancet Oncol. 2016 Dec;17(12):1653-1660. doi: 10.1016/S1470-2045(16)30562-9. Epub 2016 Nov 4. PMID 27825636
- [Derived] Wu H, Shih JY, Yang JC. Rapid Response to Sunitinib in a Patient with Lung Adenocarcinoma Harboring KIF5B-RET Fusion Gene. J Thorac Oncol. 2015 Sep;10(9):e95-e96. doi: 10.1097/JTO.0000000000000611. No abstract available. PMID 26291023
- [Derived] Drilon A, Wang L, Hasanovic A, Suehara Y, Lipson D, Stephens P, Ross J, Miller V, Ginsberg M, Zakowski MF, Kris MG, Ladanyi M, Rizvi N. Response to Cabozantinib in patients with RET fusion-positive lung adenocarcinomas. Cancer Discov. 2013 Jun;3(6):630-5. doi: 10.1158/2159-8290.CD-13-0035. Epub 2013 Mar 26. PMID 23533264
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/